CLINICAL TRIAL: NCT03955939
Title: A Phase 1b Study of Aurora A Kinase Inhibitor LY3295668 Erbumine in Monotherapy and Combination Therapy in Patients With Metastatic Breast Cancer Post CDK4/6 Inhibitor and Endocrine Therapy
Brief Title: A Study of LY3295668 Erbumine in Participants With Breast Cancer That Has Spread to Other Parts of the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17249; J1O-MC-JZHC (Other: Eli Lilly and Company); 2018-004183-61 (EudraCT Number)
Record Dates: First submitted 2019-05-17; First posted 2019-05-20 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Metastatic Breast Cancer
Keywords: aurora kinase A; kinase; aurora A; aurora kinase inhibitor; aurora kinase A inhibitor; kinase inhibitor; AURKA; AurA
MeSH Terms: conditions — Breast Neoplasms; Epilepsy | interventions — LY3295668 erbumine; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- LY3295668 Erbumine Part A (Experimental): LY3295668 erbumine administered orally (Part I).
  Approximately the first 10 participants enrolled in this arm will be administered midazolam.
  Interventions: Drug: LY3295668 Erbumine; Drug: Midazolam
- LY3295668 Erbumine Part B (Experimental): LY3295668 erbumine administered orally (Part I).
  Approximately the first 10 participants enrolled in this arm will be administered midazolam.
  Interventions: Drug: LY3295668 Erbumine; Drug: Midazolam
- LY3295668 Erbumine + Endocrine Therapy Cohort 1 (Experimental): LY3295668 erbumine administered orally and endocrine therapy administered according to package label (Part II).
  Interventions: Drug: LY3295668 Erbumine; Drug: Endocrine therapy
- LY3295668 Erbumine + Endocrine Therapy Continuation Part C (Experimental): LY3295668 erbumine administered orally and endocrine therapy administered according to package label (Part I).
  Interventions: Drug: LY3295668 Erbumine; Drug: Endocrine therapy
- LY3295668 Erbumine + Endocrine Therapy Switch Part D (Experimental): LY3295668 erbumine administered orally and endocrine therapy administered according to package label (Part I).
  Interventions: Drug: LY3295668 Erbumine; Drug: Endocrine therapy

INTERVENTIONS:
Drug: LY3295668 Erbumine — Administered orally.
Drug: Endocrine therapy — Administered according to label instructions.
  Arms: LY3295668 Erbumine + Endocrine Therapy Cohort 1; LY3295668 Erbumine + Endocrine Therapy Continuation Part C; LY3295668 Erbumine + Endocrine Therapy Switch Part D
Drug: Midazolam — Administered orally.
  Arms: LY3295668 Erbumine Part A; LY3295668 Erbumine Part B

SUMMARY:
The reason for this study is to determine the recommended phase 2 dose of the study drug LY3295668 erbumine in participants with breast cancer that has spread to other parts of the body.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have hormone receptor positive and HER2 negative metastatic breast cancer
* Participant must have progressed on at least 1 line of endocrine therapy and 1 cyclin dependent kinase (CDK)4/6 inhibitor
* Participant must be able and willing to undergo mandatory tumor biopsy
* Participant must have normal organ function
* Participant must be able to swallow capsules

Exclusion Criteria:

* Participant must not have had prior chemotherapy for mBC. Chemotherapy in the adjuvant/neoadjuvant setting is permitted
* Participant must not be currently enrolled in a clinical study
* Participant must not have another serious medical condition
* Participant must not have previously received an aurora kinase inhibitor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Reductions | Baseline through Cycle 1 (28 Day Cycle)
  Number of Participants with Dose Reductions
Part II: Number of Participants with Dose Limiting Toxicities (DLTs) | Baseline through Cycle 1 (28 Day Cycle)
  Part II: Number of Participants with DLTs
Overall Response Rate (ORR): Percentage of Participants Who Achieve Complete Response (CR) or Partial Response (PR) | Baseline through Measured Progressive Disease (Estimated up to 23 Months)
  ORR
Duration of Response (DoR) | Date of CR or PR to Date of Disease Progression or Death Due to Any Cause (Estimated up to 23 Months)
  DoR

SECONDARY OUTCOMES:
Clinical Benefit Rate (CBR): Percentage of Participants Who Achieve CR, PR or SD With a Duration of At Least 6 Months | Baseline through Disease Progression or Death Due to Any Cause (Estimated up to 23 Months)
  CBR
Progression-Free Survival (PFS) | Baseline to Objective Progression or Death Due to Any Cause (Estimated up to 23 Months)
  PFS
Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC) of LY3295668 | Predose Cycle 1 Day 1 through Cycle 2 Day 1 (28 Day Cycles)
  PK: AUC of LY3295668
PK: AUC of LY3295668 in Combination with Endocrine Therapy | Predose Cycle 1 Day 1 through Cycle 2 Day 1 (28 Day Cycles)
  PK: AUC of LY3295668 in Combination with Endocrine Therapy
PK: AUC of Endocrine Therapy in Combination with LY3295668 | Predose Cycle 1 Day 1 through Cycle 2 Day 1 (28 Day Cycles)
  PK: AUC of Endocrine Therapy in Combination with LY3295668
PK: AUC of Midazolam | Predose Cycle 1 Day 1 through Cycle 2 Day 1 (28 Day Cycles)
  PK: AUC of Midazolam
PK: AUC of Midazolam in Combination with LY3295668 | Predose Cycle 1 Day 1 through Cycle 2 Day 1 (28 Day Cycles)
  PK: AUC of Midazolam in Combination with LY3295668

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- United States (3):
  - City of Hope National Medical Center, Duarte, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
- Belgium (4):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3295668 Erbumine in Participants With Breast Cancer That Has Spread to Other Parts of the Body — https://www.lillytrialguide.com/en-US/studies/metastatic-breast-cancer/JZHC